CLINICAL TRIAL: NCT06321172
Title: Preliminary Evaluation of the Effectiveness of FES Cycling in Terms of Training Performance, Morpho-functional Characteristics of the Leg Muscles and Bone Trophism After 6 Months of Training in Spinal Cord Injury Subjects
Brief Title: Muscle and Bone Changes After 6 Months of FES Cycling
Acronym: FES-Bike
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Eugenio Medea (Other)
Collaborators: Politecnico di Milano (Other); Villa Beretta Rehabilitation Center (Other); National Research Council (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 785
Record Dates: First submitted 2024-03-14; First posted 2024-03-20 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Spinal Cord Injuries
Keywords: Spinal Cord Injury; FES; FES cycling
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- FES cycling group (Experimental): Six months of FES-cycling trainings twice a week were performed for each pilot. Each session includes at most 30 minutes of stimulation.
  Interventions: Device: FES Bike

INTERVENTIONS:
Device: FES Bike — Six months of FES-cycling trainings twice a week is performed for each pilot. Each session includes at most 30 minutes of stimulation. At the beginning of the training period, a conditioning phase is performed until the pilot reaches pedalling autonomy. This period is also used to define the stimulation parameters (minimum and maximum values of current intensity and pulse width), reference cadence and gear, specific for the ability of each pilot. Then the training period starts and is performed indoor, setting the resistance of the smart trainer at 10% for all the participants. The sessions are organized as follows: a 3-minute warmup followed by four sets of 6 minutes of pedalling and a 3-minute cool down.

SUMMARY:
The goal of this clinical trial is to assess the effectiveness of FES cycling in terms of changes morpho-functional characteristics of the leg muscles, training performance and bone trophism in 5 subjects with Spinal Cord Injury after 6 months of training. The main question[s] it aims to answer are:

* Do the morpho-functional characteristics of the leg muscles improve after 3 and 6 months of training with FES cycling? If any, the morpho-functional improvements are maintained one month after the end of the training?
* Does the quality of the leg bones improve after 3 and 6 months of training with FES cycling?
* Does the training performance improve during the training with FES cycling?
* Do the data referred to the vegetative nervous system change after 3 and 6 months of training with FES cycling? If yes, the changes in the vegetative nervous system are maintained one month after the end of the training?
* Does the intestinal function change after 3 and 6 months of training with FES cycling? If yes, the changes are maintained one month after the end of the training?
* Does the level of spasticity of the lower limbs change after 3 and 6 months of training with FES cycling? If yes, the changes are maintained one month after the end of the training?
* Does the level of pain perceived by pilots change after 3 and 6 months of training with FES cycling? If yes, the changes are maintained one month after the end of the training?
* Does the Psychological General Well-Being of the pilots change after 3 and 6 months of training with FES cycling? If yes, the changes are maintained one month after the end of the training?
* Does the pilots' motivation in carrying out a sporting activity change between T1 (3 months after starting the training) and T2(6 months after starting the training)?

Participants will train for 6 months with FES-cycling twice a week. Each session includes at most 30 minutes of stimulation.

DETAILED DESCRIPTION:
Six months of FES-cycling trainings twice a week is performed for each pilot. Each session includes at most 30 minutes of stimulation.

At the beginning of training period, a conditioning phase is performed until the pilot reaches pedalling autonomy. This period is also used to define the stimulation parameters (minimum and maximum values of current intensity and pulse width), reference cadence and gear, specific for the ability of each pilot. Then the training period start and is performed indoor, setting the resistance of the smart trainer at 10% for all the participants. The sessions are organized as follows: a 3-minute warmup followed by four sets of 6 minutes of pedalling and a 3-minute cool down.

ELIGIBILITY:
Inclusion Criteria:

* Age of subjects between 18 and 65 years.
* Subjects with paraplegia resulting from a SCI with both traumatic and non-traumatic origins occurred less than 5 years before the start of the study.
* Complete loss of motor function in the lower limbs (level ≤ T3, American Spinal Injury Association (ASIA) scale A or B)
* Adequate control of the trunk and sufficient muscle contraction using FES with surface electrodes.
* Preference for subjects with an aptitude for sports practice.
* Absence of a level of spasticity preventing device use and of disabling pain during training

Exclusion Criteria:

* Critical osteoporosis
* Skin lesions in interfaces parts with the trike,
* Dysfunction of the autonomic nervous system, and
* Psychopathological comorbidities

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2022-09-09 (Actual); Primary Completion 2024-01-22 (Actual); Study Completion 2024-04-29 (Actual)

PRIMARY OUTCOMES:
Changes in the morpho-functional characteristics of the thigh muscles of the dominant limb | After 6 months of training
  The primary outcome is the changes in the morpho-functional characteristics of the thigh muscles of the dominant limb, which is investigated with the Magnetic Resonance Imaging (MRI) with multiparametric investigation methods.

SECONDARY OUTCOMES:
Changes in the morpho-functional characteristics of the thigh muscles of the dominant limb | After 3 months of training
  The primary outcome is the changes in the morpho-functional characteristics of the thigh muscles of the dominant limb, which is investigated with the Magnetic Resonance Imaging (MRI) with multiparametric investigation methods.
Changes in the morpho-functional characteristics of the thigh muscles of the dominant limb | One month after the end of the training
  The primary outcome is the changes in the morpho-functional characteristics of the thigh muscles of the dominant limb, which is investigated with the Magnetic Resonance Imaging (MRI) with multiparametric investigation methods.
Changes in bone quality | After 6 months of training
  The evaluation of improvements in the quality of the leg bones is performed with the Bone Mineral Density (BMD)
Changes in data referring to the vegetative nervous system | After 3 months of training
  The evaluation of vegetative nervous system includes a series of test: at the beginning a rest test, then a standing test and a stepping test using a step automatic induction system (Erigo, Hocoma) and finally a cycling test (LAMBDA). For all these tests, heart rate (HR), systolic and diastolic blood pressure (sBP and dBP) and total peripheral resistance index (TPRI) are recorded.
Changes in data referring to the vegetative nervous system | After 6 months of training
  The evaluation of vegetative nervous system includes a series of test: at the beginning a rest test, then a standing test and a stepping test using a step automatic induction system (Erigo, Hocoma) and finally a cycling test (LAMBDA). For all these tests, heart rate (HR), systolic and diastolic blood pressure (sBP and dBP) and total peripheral resistance index (TPRI) are recorded.
Changes in data referring to the vegetative nervous system | One month after the end of the training
  The evaluation of vegetative nervous system includes a series of test: at the beginning a rest test, then a standing test and a stepping test using a step automatic induction system (Erigo, Hocoma) and finally a cycling test (LAMBDA). For all these tests, heart rate (HR), systolic and diastolic blood pressure (sBP and dBP) and total peripheral resistance index (TPRI) are recorded.
Changes in the intestinal function | After 3 months of training
  Neurogenic Bowel Dysfunction (NBD) score is used to evaluate intestinal function.
Changes in the intestinal function | After 6 months of training
  Neurogenic Bowel Dysfunction (NBD) score is used to evaluate intestinal function.
Changes in the intestinal function | One month after the end of the training
  Neurogenic Bowel Dysfunction (NBD) score is used to evaluate intestinal function.
Changes in the level of spasticity of the lower limbs | After 3 months of training
  To determine the level of spasticity in the lower limbs the Modified Ashworth scale (MAS) is used.
Changes in the level of spasticity of the lower limbs | After 6 months of training
  To determine the level of spasticity in the lower limbs the Modified Ashworth scale (MAS) is used.
Changes in the level of spasticity of the lower limbs | One month after the end of the training
  To determine the level of spasticity in the lower limbs the Modified Ashworth scale (MAS) is used.
Changes in the level of pain perceived | After 3 months of training
  Numerical Rating Scale (NRS) to quantify the level of pain perceived by the subject.
Changes in the level of pain perceived | After 6 months of training
  Numerical Rating Scale (NRS) to quantify the level of pain perceived by the subject.
Changes in the level of pain perceived | One month after the end of the training
  Numerical Rating Scale (NRS) to quantify the level of pain perceived by the subject.
Changes in the General Well Being of the pilots while training | After 3 months of training
  Psychological General Well-Being Index (PGWBI) is used to evaluate any repercussions that continuous FES-cycling activity has carried out on the well-being of the participants.
Changes in the General Well Being of the pilots while training | After 6 months of training
  Psychological General Well-Being Index (PGWBI) is used to evaluate any repercussions that continuous FES-cycling activity has carried out on the well-being of the participants.
Changes in the General Well Being of the pilots while training | One month after the end of the training
  Psychological General Well-Being Index (PGWBI) is used to evaluate any repercussions that continuous FES-cycling activity has carried out on the well-being of the participants.
Pilots' motivation in carrying out a sporting activity | After 3 months of training
  Sport Motivation Scale questionnaire is administered to evaluate the drivers' motivation in carrying out a sporting activity.
Pilots' motivation in carrying out a sporting activity | After 6 months of training
  Sport Motivation Scale questionnaire is administered to evaluate the drivers' motivation in carrying out a sporting activity.

CONTACTS AND LOCATIONS:
Locations (1):
- Scientific Institute, IRCCS E. Medea, Bosisio Parini, Lecco, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Sanna N, Nossa R, Biffi E, Guanziroli E, Diella E, Ferrante S, Molteni F, Peruzzo D, Casali N, Mastropietro A, Rizzo G, Tarabini M, Pedrocchi A, Ambrosini E. Evaluating the health and fitness benefits of a 6-month FES-cycling program on a recumbent trike for individuals with motor complete SCI: a pilot study. J Neuroeng Rehabil. 2025 Mar 10;22(1):55. doi: 10.1186/s12984-025-01585-0. PMID 40065341